CLINICAL TRIAL: NCT01692184
Title: A Phase 1, Two-part Study to Investigate the Safety and Pharmacokinetics of AVL-292 Following Multiple Oral Doses and to Evaluate the Effect of Food on the Pharmacokinetics of AVL-292 Following a Single Oral Dose in Healthy Adult Subjects
Brief Title: Safety and Pharmacokinetics of AVL-292 Following Multiple Doses and the Effect of Food on the Single-dose Pharmacokinetics of AVL-292
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AVL-292-004
Record Dates: First submitted 2012-09-21; First posted 2012-09-25 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Healthy
Keywords: AVL-292; Safety; Pharmacokinetics; Pharmacodynamics; Pharmacology, Clinical

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- 50 mg of AVL-292 and Placebo (Experimental): 50 mg AVL-292 (2 x 25 mg AVL-292 capsules and 6 placebo capsules) once daily for 7 days administered orally under fasted condition
  Interventions: Drug: 50 mg AVL-292; Drug: Placebo capsules
- 100 mg of AVL-292 and Placebo (Experimental): 100 mg AVL-292 (4 x 25 mg AVL-292 capsules and 4 placebo capsules) once daily for 7 days administered orally under fasted condition
  Interventions: Drug: 100 mg AVL-292; Drug: Placebo capsules
- 200 mg AVL-292 (Experimental): 8 x 25 mg AVL-292 capsules orally once daily for 7 days under fasted condition
  Interventions: Drug: 200 mg AVL-292
- 350 mg of AVL-292 (Experimental): 350 mg AVL-292 (14 x 25 mg AVL-292 capsules) once daily for 7 days administered orally under fasted condition
  Interventions: Drug: 350 mg AVL-292
- Placebo - 8 capsules (Placebo Comparator): 8 placebo capsules once daily for 7 days administered orally under fasted condition
  Interventions: Drug: Placebo capsules
- Placebo - 14 capsules (Placebo Comparator): 14 placebo capsules once daily for 7 days administered orally under fasted condition
  Interventions: Drug: Placebo capsules

INTERVENTIONS:
Drug: 50 mg AVL-292
  Other Names: AVL-292
  Arms: 50 mg of AVL-292 and Placebo
Drug: 100 mg AVL-292
  Other Names: AVL-292
  Arms: 100 mg of AVL-292 and Placebo
Drug: 200 mg AVL-292
  Other Names: AVL-292
  Arms: 200 mg AVL-292
Drug: 350 mg AVL-292
  Other Names: AVL-292
  Arms: 350 mg of AVL-292
Drug: Placebo capsules
  Arms: 100 mg of AVL-292 and Placebo; 50 mg of AVL-292 and Placebo; Placebo - 14 capsules; Placebo - 8 capsules

SUMMARY:
This is a 2-part study. The first part is to evaluate the safety, pharmacokinetics (PK) and pharmacodynamics of AVL-292 following multiple oral doses; and the second part is to evaluate the effect of food on the pharmacokinetics of a single oral dose of AVL-292.

DETAILED DESCRIPTION:
Part 2 is an open-label, randomized, 2-period, 2-way crossover study to evaluate the effect of a standard high-fat breakfast on the pharmacokinetics of AVL-292. Ten subjects will be enrolled to receive 2 single doses of 200 mg AVL-292, one with food (i.e., fed) and the other without (i.e., fasted), in a randomized sequence.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects of any ethnic origin between ages of 18 and 65 with a body mass index between 18 and 33

Exclusion Criteria:

* Recent history (i.e., within 3 years) of any clinically significant neurological, gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, endocrine, hematological, dermatological, psychological, ophthalmological, allergic or other major disorders;
* Use of any prescribed systemic or topical medication within 30 days of the first dose;
* Use of any non-prescribed systemic or topical medication (including vitamin/mineral supplements and herbal medicines, e.g., St. John's Wort) within 7 days of the first dose administration;
* Exposure to an investigational drug (new chemical entity) within 30 days prior to the first dose administration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2012-08-01 (Actual); Primary Completion 2012-10-08 (Actual); Study Completion 2012-10-08 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Up to 28 days after last AVL-292 dose
  Number of participants with adverse events
PK-(Cmax) | 24 hours after the last AVL-292 dose on days 1 and 7
  Maximum observed concentration in plasma
PK-(AUC) | 24 hours after the last AVL-292 dose days 1 and 7
  Area under the plasma concentration-time curve

SECONDARY OUTCOMES:
Pharmacodynamic response measured in percentage of target occupancy by AVL-292 in peripheral blood mononuclear cells | 24 hours after the last AVL-292 dose days 1 and 7
  Pharmacodynamic response measured in percentage of target occupancy by AVL-292 in peripheral blood mononuclear cells

CONTACTS AND LOCATIONS:
Overall Officials: Maria Palmisano, MD, Study Director — Celgene Corporation
Locations (1):
- Covance Clinical Research Unit, Dallas, Texas, United States